CLINICAL TRIAL: NCT06302829
Title: Comparison of Intramuscular Electrical Stimulation Versus Dry Needling on Active Trigger Points of Adhesive Capsulitis
Brief Title: Comparison of IMES Versus DN on ATrPs of AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Shafia Anjum
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Shoulder Pain
Keywords: trigger points; range of motion; dry needling; disability
MeSH Terms: conditions — Shoulder Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Masking Description: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramuscular Electrical stimulation (Experimental): Myofascial trigger point would be targeted by direct intramuscular electrical stimulation by using direct electrode placement method, where anode pole and the cathode pole of the stimulator connected to the needles of the MTrPs of the shoulder girdle muscles using the alligator clip connector in which both electrodes are on the muscle belly in which anode pole at proximal end and cathode pole at the distal end along the musculotendinous junction. The special programmed comfy stim (a double channeled multipurpose electrical stimulator) was used to deliver electrical impulses with following parameters; pulse duration 80µs, frequency 100HZ, and time duration for 10 min
  Interventions: Other: intramusuar electrical stimulation
- Dry Needling (Active Comparator): DN for the MTrPs will be performed over the identified trigger points locations at a suitable angle. The needles of suitable length and thickness (30-mm), depending on the depth of the MTrPs location inserted into the shoulder girdle muscles to deactivate the active MTrPs. Subsequently, the inserted needles moved to-and-fro direction to elicit the local twitch responses, which further reaffirms the ideal placement of needle into the MTrPs. After the twitch response obtained, the dry needles were kept within the muscles approximately for 10 minutes. Dry needling was performed subscapularis, latissimus dorsi, supraspinatus, deltoid, teres minor.
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Dry needling — AROM 10 repetitions ×2 set×30 sec ,6days\week, Shoulder strengthening exercises: Isometric pain free (elastic Thera-band) 10 repetitions ×2 set×30 sec ,6days\week, Maitland mobilization grade 3 and 4 10 repetitions ×2 set×30 sec ,6days\week Total of 6 session were given each consisting of 30min
  Other Names: conventional treatment
  Arms: Dry Needling
Other: intramusuar electrical stimulation — Myofascial trigger point would be targeted by direct intramuscular electrical stimulation by using direct electrode placement method, where anode pole and the cathode pole of the stimulator connected to the needles of the MTrPs of the shoulder girdle muscles .AROM 10 repetitions ×2 set×30 sec ,6days\week, Shoulder strengthening exercises: Isometric pain free (elastic Thera-band) 10 repetitions ×2 set×30 sec ,6days\week, Maitland mobilization grade 3 and 4 10 repetitions ×2 set×30 sec ,6days\week Total of 6 session were given each consisting of 30 min
  Other Names: conventional treatment
  Arms: Intramuscular Electrical stimulation

SUMMARY:
The aim of our study to compare DN and IMES for pressure pain threshold, ROM and the shoulder function in active trigger points with adhesive capsulitis. This study will add to the growing body of knowledge that if these two techniques yield comparable outcomes and if one technique is superior to the other, which should be the alternative of therapy. Moreover, it would add to the society as there are very limited researches done in Pakistan using needling for trigger points in adhesive capsulitis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 60 year of both genders
* Diagnosed patients of stage 3 Adhesive capsulitis with type I and II diabetes
* Involvement of at least 3 shoulder girdle muscles in Active MTrPs (subscapularis, latissimus dorsi, deltoid (anterior, middle, posterior)
* Active MTrPs in shoulder girdle muscles (subscapularis, supraspinatus, deltoid (anterior, middle, posterior), teres minor, latissimus dorsi)
* Reproduction of the patient's symptoms at active trigger point, Taut band, Hypersensitive spot, Referred pain pattern, local twitch response
* Minimum 60 degrees of active/passive shoulder abduction range of movement.

Exclusion Criteria:

* Systemic inflammatory joint disease of shoulder joint (RA, OA polymyalgia rheumatic)
* Cerebral Vascular Accident
* Fibromyalgia, neurological deficits of upper limb (Nerve root entrapment, Cervical radiculopathy, Thoracic outlet syndrome)
* History of Fracture, Dislocation, Acute soft tissue injury, Acute bursitis
* Avascular necrosis of humeral head or visceral referred pain to shoulder
* Pregnancy, Hypothyroidism, skin infection
* Patients who are using Antiplatelet Therapy with in past 3 days of study
* Extreme fear of needles

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2024-01-21 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Algometer (pressure pain threshold) | 3rd week
  This tool can be used to assess the participant pressure pain at baseline ,2nd week,3rd week post assessment. Pressure pain threshold is measured at active trigger point at subscapularis, deltoid (ant, middle, post), latissimus dorsi, teres minor, supraspinatus. The PPT are measured by mean and standard deviation kg\cm2

SECONDARY OUTCOMES:
ROM Shoulder (Flexion) | 3rd week
  Changes from baseline,2nd week,3rd week ROM range of motion of shoulder flexion was taken
ROM Shoulder (Abduction) | 3rd week
  Changes from baseline,2nd week,3rd week ROM range of motion of shoulder abduction was taken
ROM Shoulder (External rotation) | 3rd week
  Changes from baseline,2nd week,3rd week ROM range of motion of shoulder External rotation was taken with the help of Digital Goniometer
ROM Shoulder (Internal Rotation) | 3rd week
  Changes from baseline,2nd week,3rd week ROM range of motion of shoulder Internal rotation was taken with the help of Digital Goniometer
American shoulder and elbow surgeons scale | 3rd week
  Changes from baseline,2nd week,3rd week, American shoulder and elbow surgeons scale (ASES) Scale scoring was done at 2 level, pain questionnaire 5× (10-Q7 value), ADL Questionnaire (5× (raw score) divided by 3, final scoring is done by adding pain score and ADL score. A total 100-point scale Minimum score 0 which mean worst shoulder function and maximum score 100 which mean better shoulder function.

CONTACTS AND LOCATIONS:
Overall Officials: Aneela zia, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Railway general hopsital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No